CLINICAL TRIAL: NCT04766762
Title: A Randomized Controlled Trial of Acupuncture in Treating Migraine Without Aura by the Method of Regulating Ying and Wei
Brief Title: A Randomized Controlled Trial of Acupuncture in Treating Migraine
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: The Third Affiliated hospital of Zhejiang Chinese Medical University (Other)
Responsible Party: Principal Investigator, Chuanlong Zhou, Deputy chief physician of TCM, The Third Affiliated hospital of Zhejiang Chinese Medical University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2020ZB125
Record Dates: First submitted 2021-02-17; First posted 2021-02-23 (Actual); Last update posted 2022-07-11 (Actual); Status verified 2022-07

CONDITIONS: Migraine Without Aura
Keywords: migraine, acupuncture, randomized controlled trial
MeSH Terms: conditions — Migraine without Aura; Migraine Disorders | interventions — Flunarizine

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Acupuncture combined with placebo group (Experimental): Patients in this group will receive acupuncture combined with placebo.
  Interventions: Procedure: Acupuncture combined with placebo
- Sham acupuncture combined with medication group (Other): Participants in this group will receive sham acupuncture plus flunarizine hydrochloride.
  Interventions: Procedure: Sham acupuncture combined with flunarizine hydrochloride

INTERVENTIONS:
Procedure: Acupuncture combined with placebo — This group will include 48 patients. Patients in this group will receive acupuncture combined with placebo. Participants are in the supine position. The bilateral Tianrong (SI 17) acupoints are needled for 1-1.5 inch with the direction tilted back 45±5 degrees. The bilateral Fengchi (GB 20) acupoints are needled for 0.5-1 inch with the direction tilted to nose. The bilateral Neiguan (PC 6) acupoints are also needled for 0.5-1 inch with the straight direction. In addition, 4-6 additional acupoints can be identified according to different syndrome types of patients. The needles are kept for 30 min, the treatment frequency is 3 times per week, and the treatment duration lasts 8 weeks. Meanwhile, the dosage of placebo is 1 capsule twice a day and the treatment duration also lasts 8 weeks.
  Arms: Acupuncture combined with placebo group
Procedure: Sham acupuncture combined with flunarizine hydrochloride — This group will include 48 patients. Participants in this group will receive sham acupuncture plus flunarizine hydrochloride. Participants are in the supine position and sham acupuncture is conducted. The bilateral Tianrong (SI 17) acupoints, Fengchi (GB 20) acupoints and Neiguan (PC 6) acupoints are selected, and 4-6 additional acupoints can be identified according to the syndrome type of the participants. The needles are kept for 30 min, the treatment frequency is 3 times per week, and the treatment duration lasts 8 weeks. Moreover, the dosage of flunarizine hydrochloride is 5mg twice a day and the treatment duration also lasts 8 weeks.
  Arms: Sham acupuncture combined with medication group

SUMMARY:
Migraine without aura is a common kind of nervous system diseases that can easily cause recurrent headache, leading to severe impacts on quality of life and health care costs. Current therapeutic options for migraine without aura mainly include flunarizine hydrochloride that can relieve vasospasm. Nevertheless, the efficacy of flunarizine hydrochloride is always limited by inevitable side effects, which result in poor compliance of patients. Moreover, for some most suffering patients, the control of pain is often unsatisfactory despite of the administration of complex treatment combinations.

As a non-pharmaceutical therapy, acupuncture is widely used for a wide range of pain conditions. Thus, it might be an alternative treatment for migraine without aura. The aim of this randomized controlled trial is to investigate the efficacy and safety of acupuncture therapy in patients with migraine without aura from the perspective of Regulating Ying and Wei.

DETAILED DESCRIPTION:
This randomized controlled trial will enroll 96 migraine patients without aura from the Third Affiliated Hospital of Zhejiang Chinese Medical University. All patients will be randomly assigned to either the acupuncture combined with placebo group or sham acupuncture combined with medication group through a randomization system. Primary outcome will be pain intensity assessed by visual analogue scale (VAS) scale. Secondary outcomes will include migraine-specific quality of life (MSQOL) scale and headache needs assessment survey (HANA) questionnaire scale.

ELIGIBILITY:
Inclusion Criteria:

1. Patients meet the diagnostic criteria of migraine without aura;
2. 25 ≤ age ≤50 years, male or female;
3. The efficacy of drugs and other therapeutic methods is not obvious; the frequency of migraine attacks in the past 3 months is more than twice a month;
4. Drug treatment for migraine without aura is stopped for at least one week;
5. Participants can understand the study protocol and written informed consent is signed.

Exclusion Criteria:

1. Patients have severe complications in cardiovascular, liver, kidney, hematopoietic and other systems;
2. Pregnant or lactating women;
3. Patients have spontaneous bleeding tendency so it is not suitable for them to receive acupuncture;
4. Patients have an allergic history of flunarizine hydrochloride or a history of depression;
5. Patients are diagnosed as psychosis.

Ages: 25 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 96 (Estimated)
Dates: Start 2021-04-21 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-02-28 (Estimated)

PRIMARY OUTCOMES:
Change in pain intensity | Baseline，4 weeks after treatment，8 weeks after treatment，4 weeks after follow-up visiting，12 weeks after follow-up visiting，and 24 weeks after follow-up visiting
  Change in Pain intensity will be measured by visual analog scale (VAS)，he VAS divides the pain from 0 to 10 into 11 grades. 0: No pain; 10: the worst pain; ≤3: mild pain; 4-6: moderate pain which is tolerable; 7-10: severe pain which is unbearable.
Change in number of migraine attacks per 4 weeks | Baseline，4 weeks after treatment，8 weeks after treatment，4 weeks after follow-up visiting，12 weeks after follow-up visiting，and 24 weeks after follow-up visiting
  Change in Number of migraine attacks is assessed by patients' pain diary

SECONDARY OUTCOMES:
Migraine-specific Quality of life | Baseline，4 weeks after treatment，8 weeks after treatment，4 weeks after follow-up visiting，12 weeks after follow-up visiting，and 24 weeks after follow-up visiting
  Quality of life will be measure by migraine-specific quality of life (MSQOL) scale.This questionnaire consists of 25 items, with 4 answers for each question. The overall format and scores are as follows: 1.Very much; 2. Many; 3. Some; 4. Not at all. The overall scale ranges from 25 to 100, with higher scores indicating the better quality of life.
Headache Needs Assessment Survey (HANA) Questionnaire Scale | Baseline，4 weeks after treatment，8 weeks after treatment，4 weeks after follow-up visiting，12 weeks after follow-up visiting，and 24 weeks after follow-up visiting
  Evaluate the frequency and severity of the migraine effect.The overall score ranges from 14 to 70, with higher scores indicating the greater impact of migraine on life.

CONTACTS AND LOCATIONS:
Overall Officials: Chuanlong Zhou, Principal Investigator — The Third Affiliated hospital of Zhejiang Chinese Medical University
Locations (1):
- The Third Affiliated Hospital of Zhejiang Chinese Medical University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Zhou C, Bao J, Hu H, Ye S, Shao X, Liang Y, Fang J. Acupuncture Based on Regulating Autonomic Nerves for the Prevention of Migraine Without Aura: A Prospective, Double-Dummy, Randomized Controlled Clinical Trial. J Pain Res. 2022 Aug 4;15:2211-2221. doi: 10.2147/JPR.S372311. eCollection 2022. PMID 35957963